CLINICAL TRIAL: NCT01870596
Title: Randomized Phase II Trial of Timed Sequential Cytosine Arabinoside (Ara-C) With and Without the Checkpoint Kinase 1 (CHK1) Inhibitor MK-8776 in Adults With Relapsed AML
Brief Title: Cytarabine With or Without SCH 900776 in Treating Adult Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01097; NCI-2013-01097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); J1319 (Other: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital); 9362 (Other: CTEP); U01CA070095 (NIH); P30CA006973 (NIH)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: Adult Acute Megakaryoblastic Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With Minimal Differentiation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Adult Erythroleukemia; Adult Pure Erythroid Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute | interventions — Cytarabine; MK-8776

ARMS (2):
- Arm A (cytarabine, Chk1 inhibitor SCH 900776) (Experimental): Patients receive cytarabine IV continuously over 72 hours on days 1-3 and 10-12 and Chk1 inhibitor SCH 900776 IV over 30 minutes on days 2, 3, 11, and 12.
  Interventions: Drug: Cytarabine; Drug: CHK1 Inhibitor SCH 900776; Other: Laboratory Biomarker Analysis
- Arm B (cytarabine) (Active Comparator): Patients receive cytarabine as in Arm A.
  Interventions: Drug: Cytarabine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: CHX-3311; U-19920
Drug: CHK1 Inhibitor SCH 900776 — Given IV
  Other Names: SCH 900776
  Arms: Arm A (cytarabine, Chk1 inhibitor SCH 900776)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well cytarabine with or without SCH 900776 works in treating adult patients with relapsed acute myeloid leukemia. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or stopping them from dividing. SCH 900776 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether cytarabine is more effective with or without SCH 900776 in treating acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the rates of complete remission (CR) plus CR with incomplete recovery (CRi) achieved with cytosine arabinoside (ara-C) (cytarabine) plus the checkpoint kinase 1 (CHK1) inhibitor MK-8776 (Chk1 inhibitor SCH 900776) vs. ara-C alone for adults (ages 18-75) with relapsed acute myelogenous leukemia (AML).

SECONDARY OBJECTIVES:

I. To evaluate and compare the toxicities of ara-C + MK-8776 vs. ara-C alone. II. To determine the disease free and overall survival of those achieving response to treatment.

III. To determine the impact of MK-8776 on AML blast cell deoxyribonucleic acid (DNA) repair protein expression profiles and correlate the expression profiles with CR/CRi in response to ara-C + MK-8776 vs. ara-C alone.

IV. To evaluate and compare the amount of DNA damage induced in AML blasts by ara-C + MK-8776 vs. ara-C.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive cytarabine intravenously (IV) continuously over 72 hours on days 1-3 and 10-12 and Chk1 inhibitor SCH 900776 IV over 30 minutes on days 2, 3, 11, and 12.

ARM B: Patients receive cytarabine as in Arm A.

In both arms, courses may repeat every 28 days.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Adults with the established, pathologically confirmed diagnosis of relapsed AML
* AML that has relapsed at least once or is primary induction failure
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must be able to give informed consent
* Female patients of childbearing age must have negative pregnancy test
* Serum creatinine =< 2.0 mg/dl
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 5 x upper limit normal (ULN), unless due to Gilbert's, hemolysis or leukemic infiltration
* Alkaline phosphatase =< 5 x ULN, unless due to Gilbert's, hemolysis or leukemic infiltration
* Bilirubin =< 2.0 mg/dl, unless due to Gilbert's, hemolysis or leukemic infiltration
* Left ventricular ejection fraction >= 45% by multi gated acquisition scan (MUGA) or echocardiogram
* Baseline Fridericia corrected QT (QTcF) < 480 msec
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 30 days after study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients who have undergone stem cell transplantation (SCT), autologous or allogeneic, are eligible provided that they are >= 4 weeks from stem cell infusion, have no active graft-vs-host disease (GVHD), and meet other eligibility criteria
* Patients who fail primary induction therapy or relapse after achieving complete remission (CR) are eligible if they have undergone no more than 2 prior cytotoxic regimens (a regimen is described as a distinctive planned collection of agent[s] and/or modalities to be utilized together during a cycle or course of therapy; i.e., induction+consolidation with or without stem cell transplant [SCT]), >= 2 weeks off cytotoxic chemotherapy, and >= 2 weeks off radiation therapy; patients must be off biologic therapies including hematopoietic growth factors >= 2 weeks; if using hydroxyurea (HU), steroids, imatinib or other tyrosine kinase inhibitors (TKIs), interferon, or other non-cytotoxics for blast count control, patient must be off for >= 24 hours (hrs) before starting MK-8776
* Fluvoxamine and ciprofloxacin must be stopped 7 days prior to day 1 of therapy, and be excluded during administration of study therapy; if the subject is using any of the other drugs that are cytochrome P4501A2 (CYP1A2) or P-glycoprotein (PgP) inhibitors, substitution should be considered and administration of these drugs should be avoided on the days of administration of MK-8776; in addition, smoking should be avoided and cytochrome P450 3A4 (CYP3A4) substrates with a narrow therapeutic index should be avoided: alfentanil, astemizole, cisapride, cyclosporine, diergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, terfenadine

Exclusion Criteria:

* Any previous treatment with MK-8776
* Considered refractory or treatment failure to most recent treatment regimen, unless primary refractory
* Concomitant chemotherapy, radiation therapy, or immunotherapy
* Hyperleukocytosis with >= 50,000 blasts/uL (if using HU, steroids, tyrosine kinase/src inhibitors (including fms-related tyrosine kinase 3 [FLT3] inhibitors), arsenic, interferon or leukapheresis for blast count control, patient must be off those agents for 24 hours prior to beginning ara-C +/- MK-8776)
* Acute progranulocytic leukemia (APL, M3)
* Active disseminated intravascular coagulation (DIC)
* Active central nervous system (CNS) leukemia
* Active, uncontrolled infection; patients with infection under active treatment and controlled with antibiotics are eligible
* Presence of other life-threatening illness
* Patients with mental deficits and/or psychiatric history that preclude them from giving informed consent or from following protocol
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MK-8776
* History of Fridericia corrected QT (QTcF) prolongation greater than grade 1 or 480 msec
* Subjects with the following cardiac risk factors must be excluded: transmural myocardial infarction (MI) within prior 6 months, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack (TIA) or seizure disorder within 6 months prior to study drug administration
* Subjects with history of risk factors for torsades de pointes: clinical history of heart failure (New York Heart Association [NYHA] class III or IV), hypo- or hyper-kalemia or hypomagnesemia (supplementation to bring levels within normal limits prior to administration of MK-8776 is acceptable) or family history of Long QT Syndrome
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy or who have a prior history of acquired immunodeficiency syndrome (AIDS) indicator conditions, other than history of lymphoma more than 3 years remote

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Smith, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital
Locations (5):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Cytarabine, Chk1 Inhibitor SCH 900776) | Arm B (Cytarabine)
Started | 14 | 18
Completed | 14 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Cytarabine, Chk1 Inhibitor SCH 900776) | Arm B (Cytarabine) | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 3 | 6 | 9
Age, Continuous [Median (Full Range); unit: years] | 60 [29 to 72] | 60 [29 to 72] | 60 [29 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Response Rate(CR/CRi) Rate
Description: For descriptive purposes, the CR/CRi (complete response/Complete response with incomplete blood count recovery) rate will be reported at the end of the study separately for Arm A and Arm B. Responses are following definitions consistent with those published by Dohner H, Estey EH, Amadori S, et al. CR is defined as Bone marrow showing less than 5% myeloblasts with normal maturation of all cell lines, an ANC of at least 1000/μL and a platelet count of 100,000/μL, absence of blasts in peripheral blood, absence of identifiable leukemic cells in the bone marrow, clearance of disease-associated cytogenetic abnormalities, and clearance of any previously existing extramedullary disease. CRi: All CR criteria except for residual neutropenia (ANC < 1000/μL)
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Arm A (Cytarabine, Chk1 Inhibitor SCH 900776) | Arm B (Cytarabine)
Number analyzed (Participants) | 14 | 18
participants | 6 | 9

ADVERSE EVENTS:
Arm/Group | Arm A (Cytarabine, Chk1 Inhibitor SCH 900776) | Arm B (Cytarabine)
Serious Adverse Events (participants affected / at risk) | 2/14 | 6/18
Other Adverse Events (participants affected / at risk) | 14/14 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Cytarabine, Chk1 Inhibitor SCH 900776) (N=14) | Arm B (Cytarabine) (N=18)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Acute Kidney Injusry (Renal and urinary disorders) | 1 (1) | 1 (1)
Cardiac arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
death multi system organ failure (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Cytarabine, Chk1 Inhibitor SCH 900776) (N=14) | Arm B (Cytarabine) (N=18)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
ADVERSE_EVENTS 9362 9362-GA079-129 1 Investigations Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
delerium (Psychiatric disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 4 (4) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
edema limbs (General disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 7 (7)
fever (General disorders) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 2 (2) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis ora (Gastrointestinal disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Phlebitis infective (Infections and infestations) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less